CLINICAL TRIAL: NCT03481829
Title: Early Tracking of Childhood Health Determinants Study
Brief Title: Early Tracking of Childhood Health Determinants (ETCHED) Study
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918071; 18-DK-N071
Record Dates: First submitted 2018-03-28; First posted 2018-03-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Diabetes Mellitus; Obesity; Fatty Liver
Keywords: American Indians, Hispanics; Obesity; Pregnancy; Diabetes; Children; Hispanics; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Children of mothers enrolled in the study
- Pregnant women and mothers: Pregnant women/mothers

SUMMARY:
Background:

Children s weight has increased sharply in recent years. This may put them at higher risk for health problems. High blood glucose in a pregnant mother and too much weight gain during pregnancy also may have long-term effects on the child s health. Children who become overweight or obese during childhood tend to remain so as adults. Researchers want to study many risk factors during and after pregnancy, and how these affect a child s development. They will also follow the mother s health and well-being after pregnancy.

Objectives:

To learn how a pregnant mother s environment, lifestyle, and health conditions may affect her child s growth and development from birth until adulthood.

Eligibility:

American Indian/Alaska Native (AI/AN) or Hispanic adult pregnant women and their offspring.

Design:

Mothers will have 3 visits during pregnancy.

In the child s first year, mothers will have 2 visits and their child will have 4.

Children will have 2 visits in their second year and 1 each year until they turn 18.

Mothers will have a visit 2 years after birth and 4-5 years later.

Both the mother and child s medical records will be reviewed. They will have physical exams and give blood and stool samples.

Mothers may give cord blood and placenta samples. They will give breastmilk and urine samples. They will fill out questionnaires.

They will have an ultrasound. They may get an activity monitor.

Mother and child will be followed until the child s 18th birthday.

DETAILED DESCRIPTION:
Study Description:

The current project will establish a longitudinal cohort of mother/infant/child dyads among American Indian/Alaska Native (AI/AN) and Hispanic ethnic groups, to study the role of a combination of biological and environmental factors on infant/childhood obesity and cardio metabolic risk.

Objectives:

Primary Objective: Primary Objective: To study the associations of maternal risk factors, including pre-pregnancy body mass index, gestational weight gain, and glycemia during pregnancy with offspring birth weight, length, and age/sex adjusted Body Mass Index (BMI) percentile and z-score up to 24-months of age.

Secondary Objectives:

1. To study the associations of maternal risk factors, including pre-pregnancy BMI, gestational weight gain, and glycemia with weight, adiposity, and physical growth patterns during childhood and adolescence (2 to 18 years of age).
2. To study the role of maternal clinical, genetic, biochemical, lifestyle, and psychosocial factors during pregnancy in mediating the associations between maternal risk factors and birth weight of the offspring, and weight, adiposity, metabolic profile, and neurodevelopment during infancy, childhood and adolescence.
3. To examine the role of family, socioeconomic, and environmental factors influencing child growth patterns, body composition and neurodevelopment in infancy and childhood.
4. To assess the frequency of hepatic steatosis in children and its association with BMI and biochemical changes
5. To examine the relationship between maternal risk factors, early childhood exposures and changes in gut microbiome during,

   infancy, childhood and adolescence.
6. To study the associations of maternal risk factors, including pre-pregnancy BMI, gestational weight gain, and glycemia and placental function, methylome, transcriptome, proteome and metabolome with weight, adiposity, and physical growth patterns during childhood and adolescence (2 to 18 years of age).

Endpoints:

Primary Endpoint: Birth weight, length, and age/sex adjusted BMI percentile and z-score up to 24-months of age (time points: 6-12

weeks, 4, 6, 12, 18, and 24 months).

Secondary Endpoints: BMI percentile and z-scores 2 years to 18 years, biochemical measures, stool microbiome, neurocognitive

development.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Pregnant women aged 18 years or older (pregnancy confirmed by urine or serum pregnancy test, or ultrasound examination)
2. American Indian or Hispanic by self-report
3. Agree to continue with research study participation (both mother and their offspring), for at least 3 years after delivery.

In case where a pregnant mother is carrying multiple fetuses (multiple pregnancy), she will be eligible to participate in this study and all her live newborns, as a result of that pregnancy, will be eligible for participation in this study. Mothers will also be eligible to participate with any consecutive pregnancies.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Women who are incarcerated or are unable to consent.
2. Women whose fetus is not viable or are not planning to continue the pregnancy.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women from the Phoenix, AZ area
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2041-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant BMI | Birth, 6 weeks, and 4, 6, 12, 18 and 24 months
  Birth weight, length, and age/sex adjusted BMI percentile and z-score up to 24-months of age (time points: 6-12 weeks, 4, 6, 12, 18 and 24 months).

SECONDARY OUTCOMES:
Child BMI | annually from age 2 to 18
  Child BMI measured annually from 2 years of age to 18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Sinha, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Genomic Data Sharing Policy, which applies to all NIH-funded research that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data.
Supporting Information: Study Protocol, ICF
Time Frame: Data from this study may be requested from other researchers 1 year after the completion of the primary endpoint by contacting the Principal Investigator.
Access Criteria: This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.

REFERENCES:
- [Background] Pettitt DJ, Aleck KA, Baird HR, Carraher MJ, Bennett PH, Knowler WC. Congenital susceptibility to NIDDM. Role of intrauterine environment. Diabetes. 1988 May;37(5):622-8. doi: 10.2337/diab.37.5.622. PMID 3360218
- [Background] Dabelea D, Hanson RL, Lindsay RS, Pettitt DJ, Imperatore G, Gabir MM, Roumain J, Bennett PH, Knowler WC. Intrauterine exposure to diabetes conveys risks for type 2 diabetes and obesity: a study of discordant sibships. Diabetes. 2000 Dec;49(12):2208-11. doi: 10.2337/diabetes.49.12.2208. PMID 11118027
- [Background] Pettitt DJ, Baird HR, Aleck KA, Bennett PH, Knowler WC. Excessive obesity in offspring of Pima Indian women with diabetes during pregnancy. N Engl J Med. 1983 Feb 3;308(5):242-5. doi: 10.1056/NEJM198302033080502. PMID 6848933
- [Derived] Arreola EV, Coonrod DV, Roy Choudhury S, Knowler WC, Hoskin M, Wasak D, Williams R, Hanson RL, Pack E, Caballero R, Gonzalez A, Sinha M. Study protocol for Early Tracking of Childhood Health determinants (ETCHED): A longitudinal observational life course study. BMC Public Health. 2024 Sep 29;24(1):2661. doi: 10.1186/s12889-024-20176-7. PMID 39343891